CLINICAL TRIAL: NCT02686138
Title: A 26-Week, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tenapanor for the Treatment of Constipation-Predominant Irritable Bowel Syndrome (IBS-C)
Brief Title: A 26-Week Study to Evaluate the Efficacy and Safety of Tenapanor in IBS-C
Acronym: T3MPO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEN-01-302
Record Dates: First submitted 2016-01-11; First posted 2016-02-19 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Constipation Predominant Irritable Bowel Syndrome
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50mg BID (Experimental): Tenapanor, 50mg BID (100mg total)
  Interventions: Drug: Tenapanor
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenapanor
  Other Names: RDX5791; AZD1722
  Arms: 50mg BID
Drug: Placebo
  Arms: Placebo

SUMMARY:
This phase 3, 26-week, randomized, double-blind, placebo-controlled, multi-center study will evaluate the safety and efficacy of one dose of Tenapanor in subjects with constipation-predominant irritable bowel syndrome (IBS-C) as defined by the ROME III criteria and who have active disease as determined after a two-week screening period. Subjects who qualify and are randomized into the study will either receive 50mg BID of Tenapanor (1:1) for a 26 week treatment period.

DETAILED DESCRIPTION:
During the 26-week double-blind treatment period, subjects will record daily assessments including: frequency and timing of bowel movements; sensation of complete bowel emptying; consistency of bowel movements; degree of straining, worst abdominal pain, abdominal discomfort, abdominal bloating, abdominal fullness and abdominal cramping; and use and timing of rescue medication. Subjects will also record weekly assessments including: adequate relief of IBS symptoms, degree of relief of IBS symptoms, IBS severity, and constipation severity.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 75 years, inclusive
* Females must be of non-childbearing potential; If of child-bearing potential, must have negative pregnancy test and confirm the use of one of the appropriate means of contraception
* Males must agree to use appropriate methods of barrier contraception or have documented surgical sterilization
* Subject meets definition of IBS-C using Rome III Criteria for the Diagnosis of IBS
* A colonoscopy based on AGA guidelines; every 10 years at ≥50 years old

Exclusion Criteria:

* Functional diarrhea as defined by Rome III criteria
* IBS with diarrhea (IBS-D), mixed IBS (IBS-M), or unsubtyped IBS as defined by Rome III criteria
* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract within 6 months prior to screening, or active disease within 6 months prior to screening; including but not limited to cancer, inflammatory bowel disease, diverticulitis, duodenal ulcer, erosive esophagitis, gastric ulcer, pancreatitis (within 12 months of screening), cholelithiasis, amyloidosis, ileus, non-controlled GERD, gastrointestinal obstruction or carcinoid syndrome.
* Potential CNS cause of constipation (e.g., Parkinson's disease, spinal cord injury, or multiple sclerosis)
* Subject has a history or current evidence of laxative abuse (in the clinical judgment of physician)
* Hepatic dysfunction (ALT [SGPT] or AST [SGOT] >2.5 times the upper limit of normal) or renal impairment (serum creatinine >2 mg/dL)
* Any evidence of or treatment of malignancy (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected) within the previous year
* Any surgery on the stomach, small intestine or colon, excluding appendectomy and cholecystectomy (unless within 60 days of screening visit)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, Ph.D., Study Chair — Ardelyx, Inc.
Locations (117):
- United States (117):
  - Ardelyx Investigative Site 257, Dothan, Alabama
  - Ardelyx Investigative Site 200, Foley, Alabama
  - Ardelyx Investigative Site 103, Huntsville, Alabama
  - Ardelyx Investigative Site 244, Huntsville, Alabama
  - Ardelyx Investigative Site 251, Huntsville, Alabama
  - Ardelyx Investigative Site 100, Huntsville, Alabama
  - Ardelyx Investigative Site 209, Saraland, Alabama
  - Ardelyx Investigative Site 210, Phoenix, Arizona
  - Ardelyx Investigative Site 296, Phoenix, Arizona
  - Ardelyx Investigative Site 269, Tucson, Arizona
  - Ardelyx Investigative Site 256, Tucson, Arizona
  - Ardelyx Investigative Site 292, Conway, Arkansas
  - Ardelyx Investigative Site 122, Little Rock, Arkansas
  - Ardelyx Investigative Site 163, Anaheim, California
  - Ardelyx Investigative Site 105, Canoga Park, California
  - Ardelyx Investigative Site 143, Chula Vista, California
  - Ardelyx Investigative Site 147, Encino, California
  - Ardelyx Investigative Site 297, La Mesa, California
  - Ardelyx Investigative Site 284, La Mirada, California
  - Ardelyx Investigative Site 107, Lomita, California
  - Ardelyx Investigative Site 165, Long Beach, California
  - Ardelyx Investigative Site 211, Orange, California
  - Ardelyx Investigative Site 233, Wheat Ridge, Colorado
  - Ardelyx Investigative Site 212, Bristol, Connecticut
  - Ardelyx Investigative Site 176, Brandon, Florida
  - Ardelyx Investigative Site 178, Cutler Bay, Florida
  - Ardelyx Investigative Site 136, Hialeah, Florida
  - Ardelyx Investigative Site 130, Hialeah, Florida
  - Ardelyx Investigative Site 191, Lynn Haven, Florida
  - Ardelyx Investigative Site 288, Miami, Florida
  - Ardelyx Investigative Site 106, Miami, Florida
  - Ardelyx Investigative Site 127, Miami Lakes, Florida
  - Ardelyx Investigative Site 179, Orlando, Florida
  - Ardelyx Investigative Site 290, Tampa, Florida
  - Ardelyx Investigative Site 254, West Palm Beach, Florida
  - Ardelyx Investigative Site 138, Atlanta, Georgia
  - Ardelyx Investigative Site 148, Atlanta, Georgia
  - Ardelyx Investigative Site 253, Atlanta, Georgia
  - Ardelyx Investigative Site 272, Decatur, Georgia
  - Ardelyx Investigative Site 229, Decatur, Georgia
  - Ardelyx Investigative Site 250, Marietta, Georgia
  - Ardelyx Investigative Site 137, Norcross, Georgia
  - Ardelyx Investigative Site 213, Savannah, Georgia
  - Ardelyx Investigative Site 124, Snellville, Georgia
  - Ardelyx Investigative Site 268, Burr Ridge, Illinois
  - Ardelyx Investigative Site 227, Evergreen Park, Illinois
  - Ardelyx Investigative Site 291, Hoffman Estates, Illinois
  - Ardelyx Investigative Site 202, Oak Lawn, Illinois
  - Ardelyx Investigative Site 218, Evansville, Indiana
  - Ardelyx Investigative Site 158, Madisonville, Kentucky
  - Ardelyx Investigative Site 270, Mandeville, Louisiana
  - Ardelyx Investigative Site 214, Marrero, Louisiana
  - Ardelyx Investigative Site 154, Metairie, Louisiana
  - Ardelyx Investigative Site 195, Shreveport, Louisiana
  - Ardelyx Investigative Site 271, Bangor, Maine
  - Ardelyx Investigative Site 160, Annapolis, Maryland
  - Ardelyx Investigative Site 255, Towson, Maryland
  - Ardelyx Investigative Site 267, Brockton, Massachusetts
  - Ardelyx Investigative Site 260, Ann Arbor, Michigan
  - Ardelyx Investigative Site 283, Buckley, Michigan
  - Ardelyx Investigative Site 239, Flint, Michigan
  - Ardelyx Investigative Site 168, Troy, Michigan
  - Ardelyx Investigative Site 216, Wyoming, Michigan
  - Ardelyx Investigative Site 221, Biloxi, Mississippi
  - Ardelyx Investigative Site 282, Jefferson City, Missouri
  - Ardelyx Investigative Site 228, St Louis, Missouri
  - Ardelyx Investigative Site 156, Billings, Montana
  - Ardelyx Investigative Site 182, Las Vegas, Nevada
  - Ardelyx Investigative Site 175, Vineland, New Jersey
  - Ardelyx Investigative Site 222, Albuquerque, New Mexico
  - Ardelyx Investigative Site 264, Albuquerque, New Mexico
  - Ardelyx Investigative Site 230, Brooklyn, New York
  - Ardelyx Investigative Site 170, Great Neck, New York
  - Ardelyx Investigative Site 203, New Hyde Park, New York
  - Ardelyx Investigative Site 205, Fayetteville, North Carolina
  - Ardelyx Investigative Site 190, Greensboro, North Carolina
  - Ardelyx Investigative Site 194, Hickory, North Carolina
  - Ardelyx Investigative Site 285, Wilmington, North Carolina
  - Ardelyx Investigative Site 172, Beavercreek, Ohio
  - Ardelyx Investigative Site 204, Cincinnati, Ohio
  - Ardelyx Investigative Site 201, Cincinnati, Ohio
  - Ardelyx Investigative Site 173, Dayton, Ohio
  - Ardelyx Investigative Site 208, Franklin, Ohio
  - Ardelyx Investigative Site 171, Huber Heights, Ohio
  - Ardelyx Investigative Site 219, Lima, Ohio
  - Ardelyx Investigative Site 232, Wadsworth, Ohio
  - Ardelyx Investigative Site 236, Oklahoma City, Oklahoma
  - Ardelyx Investigative Site 273, Tulsa, Oklahoma
  - Ardelyx Investigative Site 220, Levittown, Pennsylvania
  - Ardelyx Investigative Site 248, East Providence, Rhode Island
  - Ardelyx Investigative Site 252, Columbia, South Carolina
  - Ardelyx Investigative Site 265, Gaffney, South Carolina
  - Ardelyx Investigative Site 246, Rapid City, South Dakota
  - Ardelyx Investigative Site 261, Sioux Falls, South Dakota
  - Ardelyx Investigative Site 217, Chattanooga, Tennessee
  - Ardelyx Investigative Site 121, Franklin, Tennessee
  - Ardelyx Investigative Site 189, Hermitage, Tennessee
  - Ardelyx Investigative Site 133, Jackson, Tennessee
  - Ardelyx Investigative Site 109, Knoxville, Tennessee
  - Ardelyx Investigative Site 266, Memphis, Tennessee
  - Ardelyx Investigative Site 235, Nashville, Tennessee
  - Ardelyx Investigative Site 279, Spring Hill, Tennessee
  - Ardelyx Investigative Site 180, Channelview, Texas
  - Ardelyx Investigative Site 286, Houston, Texas
  - Ardelyx Investigative Site 262, Houston, Texas
  - Ardelyx Investigative Site 185, Houston, Texas
  - Ardelyx Investigative Site 113, McKinney, Texas
  - Ardelyx Investigative Site 263, Port Arthur, Texas
  - Ardelyx Investigative Site 181, San Antonio, Texas
  - Ardelyx Investigative Site 186, San Antonio, Texas
  - Ardelyx Investigative Site 167, Salt Lake City, Utah
  - Ardelyx Investigative Site 249, Norfolk, Virginia
  - Ardelyx Investigative Site 231, Norfolk, Virginia
  - Ardelyx Investigative Site 258, Petersburg, Virginia
  - Ardelyx Investigative Site 245, Virginia Beach, Virginia
  - Ardelyx Investigative Site 242, Spokane, Washington
  - Ardelyx Investigative Site 195, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacy BE, Shin AS, Cangemi DJ, Yang Y, Zhao S, Rosenbaum DP. Tenapanor is associated with earlier and sustained symptom relief in IBS-C: a post hoc analysis. Therap Adv Gastroenterol. 2026 Jan 24;19:17562848251414831. doi: 10.1177/17562848251414831. eCollection 2026. PMID 41601848
- [Derived] Lembo AJ, Friedenberg KA, Fogel RP, Edelstein S, Zhao S, Yang Y, Rosenbaum DP, Chey WD. Long-term safety of tenapanor in patients with irritable bowel syndrome with constipation in the T3MPO-3 study. Neurogastroenterol Motil. 2023 Nov;35(11):e14658. doi: 10.1111/nmo.14658. Epub 2023 Sep 5. PMID 37668173
- [Derived] Chey WD, Lembo AJ, Yang Y, Rosenbaum DP. Efficacy of Tenapanor in Treating Patients With Irritable Bowel Syndrome With Constipation: A 26-Week, Placebo-Controlled Phase 3 Trial (T3MPO-2). Am J Gastroenterol. 2021 Jun 1;116(6):1294-1303. doi: 10.14309/ajg.0000000000001056. PMID 33337659

RESULTS

PARTICIPANT FLOW:
Groups:
- 50mg BID: Tenapanor, 50mg BID (100mg total)
  Tenapanor
Period: Overall Study
Arm/Group | 50mg BID | Placebo
Started | 293 | 300
Completed | 219 | 235
Not Completed | 74 | 65

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50mg BID | Placebo | Total
Number analyzed (Participants) | 293 | 300 | 593
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (13.1) | 44.8 (13.8) | 45.4 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 247 | 487
  Male | 53 | 53 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 78 | 155
  Not Hispanic or Latino | 216 | 222 | 438
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 9 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 92 | 92 | 184
  White | 185 | 192 | 377
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 4 | 6
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.50 (7.18) | 30.88 (7.27) | 30.69 (7.22)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Overall Response for 6 Out of 12 Weeks
Description: An overall responder is defined as a weekly responder for the first 6/12 weeks where both CSBM and abdominal pain response criteria were met for the week. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?" The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: First 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 107 | 71
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.85

2. Secondary Outcome: Percentage of Subjects With Overall Complete Spontaneous Bowel Movement (CSBM) Response for 6 Out of 12 Weeks
Description: An overall CSBM responder is defined as a weekly responder for the first 6/12 weeks. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?"
Time Frame: First 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 139 | 100
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.11

3. Secondary Outcome: Percentage of Subjects With Overall Abdominal Pain Response for 6 Out of 12 Weeks
Description: An overall abdominal pain responder is defined as a weekly responder for the first 6/12 weeks. The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: First 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 146 | 115
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.5

4. Secondary Outcome: Percentage of Subjects With Overall Response for 13 Out of 26 Weeks
Description: An overall responder is defined as a weekly responder for the first 13/26 weeks where both CSBM and abdominal pain response criteria were met for the week. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?" The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 104 | 73
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.16

5. Secondary Outcome: Percentage of Subjects With Overall Complete Spontaneous Bowel Movement (CSBM) Response for 13 Out of 26 Weeks
Description: An overall CSBM responder is defined as a weekly responder for the first 13/26 weeks. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?"
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 121 | 93
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p = 0.01, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.3

6. Secondary Outcome: Percentage of Subjects With Overall Abdominal Pain Response for 13 Out of 26 Weeks
Description: An overall abdominal pain responder is defined as a weekly responder for the first 13/26 weeks. The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 147 | 120
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.17

7. Secondary Outcome: Percentage of Subjects With Overall Response for 9 Out of 12 Weeks
Description: An overall responder is defined as a weekly responder for the first 9/12 weeks where both CSBM and abdominal pain response criteria were met for the week. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline and a minimum of at least 3 CSBMs that same week. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?" The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: First 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 54 | 16
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.1

8. Secondary Outcome: Percentage of Subjects With Overall Complete Spontaneous Bowel Movement (CSBM) Response for 9 Out of 12 Weeks
Description: An overall CSBM responder is defined as a weekly responder for the first 9/12 weeks. The CSBM response criteria are defined as an increase of one or more change in average weekly CSBMs from baseline and a minimum of at least 3 CSBMs that same week. The definition of a CSBM is as follows: A CSBM is a spontaneous bowel movement (SBM) for which the subject responds "yes" to the following question; "Did you feel like you completely emptied your bowels?"
Time Frame: First 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 65 | 18
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.18

9. Secondary Outcome: Percentage of Subjects With Overall Abdominal Pain Response for 9 Out of 12 Weeks
Description: An overall abdominal pain responder is defined as a weekly responder for the first 9/12 weeks. The abdominal pain response criterion is defined as a decrease of 30% or more of percent change in average weekly worst abdominal pain from baseline.
Time Frame: First 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50mg BID | Placebo
Number analyzed (Participants) | 293 | 300
Participants | 105 | 80
Statistical Analysis 1: Comparison: 50mg BID vs Placebo; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.17

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 50mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/293 | 0/300
Serious Adverse Events (participants affected / at risk) | 4/293 | 8/300
Other Adverse Events (participants affected / at risk) | 47/293 | 11/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg BID (N=293) | Placebo (N=300)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
carotid artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
ovarian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
systemic inflammatory response syndrome (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50mg BID (N=293) | Placebo (N=300)
Diarrhea (Gastrointestinal disorders) | 47 (47) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT02686138/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT02686138/SAP_001.pdf